CLINICAL TRIAL: NCT04378790
Title: A Randomized Trial to Evaluate Sequential vs Simultaneous Spectacles Plus Patching for Amblyopia in Children 3 to <13 Years Old
Brief Title: A Randomized Trial to Evaluate Sequential vs Simultaneous Patching
Acronym: ATS22
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Eye Institute (NEI) (NIH); Pediatric Eye Disease Investigator Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ATS22; 2UG1EY011751 (NIH)
Record Dates: First submitted 2020-05-05; First posted 2020-05-07 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Amblyopia
Keywords: patching; glasses; spectacles; simultaneous; sequential
MeSH Terms: conditions — Amblyopia | interventions — Eyeglasses

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequential treatment (Active Comparator): full-time spectacle correction first, with subsequent patching for 2 hours per day/7 days per week only if needed (no improvement (stable/worsening) and residual)
  Interventions: Other: Patching; Other: Glasses
- Simultaneous treatment (Experimental): full-time spectacle correction and part-time patching for 2 hours per day/7 days per week
  Interventions: Other: Patching; Other: Glasses

INTERVENTIONS:
Other: Patching — Procedure in which the eye is covered utilizing a patch to increase the strength of the uncovered eye.
  Other Names: Eye Patch
Other: Glasses — Eye Glasses are created and worn by patient to improve vision
  Other Names: Spectacles

SUMMARY:
A randomized trial to determine whether simultaneous treatment with spectacles and patching has an equivalent VA outcome compared with sequential treatment, first with spectacles alone followed by patching (if needed), for previously untreated amblyopia in children 3 to <13 years of age.

DETAILED DESCRIPTION:
At an enrollment visit, distance VA will be measured in trial frames with or without cycloplegia based on a cycloplegic refraction performed within 30 days. If still apparently eligible, children will be prescribed spectacles and will then return for a spectacle baseline visit, where they will wear their new spectacles for the first time for at least 10 minutes (but no more than 24 hours) and will be tested in those new spectacles to confirm final eligibility prior to randomization.

Participants not found to be eligible in their new spectacles will end study participation. Participants eligible for the study will be randomly allocated to one of two treatment groups: Sequential (spectacles alone) and then patching if needed (monitored by ODM), or Simultaneous (spectacles and patching monitored by ODM).

After randomization, follow-up visits will occur at 8-week intervals through 56 weeks. At each visit on or after the 8-week visit, participants will be classified as either: stable/worsening or improving; those stable/worsening are then classified as having either resolved or residual amblyopia, provided that the current and most recent previous visit were completed at least 6-weeks apart (target 8 weeks) and provided the required test and retest VA testing was completed. Participants who are stable/worsening and have residual amblyopia in the sequential group will start patching (monitored by ODM) and continue to be followed every 8 weeks. Participants in the simultaneous group, or in the sequential group after having advanced to patching, who are stable/worsening but have residual amblyopia will be released to treatment at investigator discretion.

All participants continue 8-weekly visits until 56 weeks when Study participation ends.

ELIGIBILITY:
Inclusion Criteria:

1. Age 3 to <13 years at the time of randomization
2. Amblyopia associated with anisometropia, strabismus, or both

   o Criteria for strabismic amblyopia: At least one of the following must be met:
   * Presence of a heterotropia on examination at distance or near fixation (with or without optical correction)
   * Documented history of strabismus which is no longer present (which in the judgment of the investigator could have caused amblyopia)

     * Criteria for anisometropia: At least one of the following criteria must be met:

       * 1.00 D difference between eyes in spherical equivalent (SE)
       * 1.50 D difference in astigmatism between corresponding meridians in the two eyes
     * Criteria for combined-mechanism amblyopia: Both of the following criteria must be met:
   * Criteria for strabismus are met (see above)

     * 1.00 D difference between eyes in spherical equivalent OR ≥1.50 D difference in astigmatism between corresponding meridians in the two eyes
3. No previous treatment for amblyopia, including no more than 24 hours of spectacle wear.
4. Investigator planning to initiate spectacle correction of refractive error meeting the following criteria based on a cycloplegic refraction that has been performed within 30 days:

   1. Full correction of anisometropia
   2. Full correction of astigmatism with the same axis found by the cycloplegic refraction
   3. Full correction of any myopia
   4. Hyperopia must not be under corrected by more than 1.50 D, and reduction in plus sphere must be symmetric in the two eyes.
5. At enrollment, single VA measured in each eye assessed in trial frames with the spectacle correction the investigator plans to prescribe, using the investigator's routine method as follows:

   * VA in the amblyopic eye 20/40 to 20/200 inclusive.
   * Age-normal VA in the fellow eye:40,41

     * 3 years: 0.4 logMAR (20/50) or better
     * 4 years: 0.3 logMAR (20/40) or better
     * 5-6 years: 0.2 logMAR (20/32) or better
     * 7-12 years: 0.12 logMAR (78 letters) or better
   * Interocular difference ≥ 3 logMAR lines (0.3 logMAR) or ≥ 15 letters o When participants return for the Spectacle Baseline / Randomization Visit with their new spectacles, they will need to meet the same criteria as above using the ATS-HOTV or E-ETDRS protocol after wearing the new spectacles for at least 10 minutes (based upon the mean of a test and retest of VA in those new spectacles).
6. Investigator is willing to prescribe spectacle wear followed sequentially by patching or simultaneous spectacles and patching treatment per protocol.
7. Parent understands the protocol and is willing to accept randomization.
8. Parent has phone (or access to phone) and is willing to be contacted by Jaeb Center staff or other study staff.
9. Relocation outside of area of an active PEDIG site for this study within the next 56 weeks is not anticipated.

Exclusion Criteria:

1. Myopia greater than -6.00 D spherical equivalent in either eye.
2. Previous intraocular or refractive surgery.
3. Planned strabismus surgery in the next 56 weeks.
4. Any previous treatment for amblyopia (patching, atropine, Bangerter filter, vision therapy, or binocular treatment).
5. Previous spectacle or contact lens wear for more than 24 hours.
6. Parent and participant willing to forego option of contact lens wear for the duration of the study.
7. Ocular co-morbidity that may reduce VA determined by an ocular examination performed within the past 7 months (Note: nystagmus per se does not exclude the participant if the above VA criteria are met).
8. Severe developmental delay that would interfere with treatment or evaluation (in the opinion of the investigator). Participants with mild speech delay or reading and/or learning disabilities or attention deficit hyperactivity disorder (ADHD) are not excluded.
9. Known allergy to adhesive patches.
10. Known allergy to silicone.

Ages: 3 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 544 (Estimated)
Dates: Start 2020-12-08 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Mean Change in Amblyopic Eye logMAR distance Visual Acuity | 56 weeks
  1. Amblyopic eye VA (calculated as mean of test and retest) at the last visit that was the basis for a "stable resolved" or "stable residual" determination (in the sequential group, stable residual amblyopia criteria can be reached only after patching has been instituted); or
  2. 56-week visit amblyopic-eye VA (calculated as mean of test and retest) in those completing a 56-week visit without ever meeting criteria for "stable resolved" or "stable residual" amblyopia (if retest missing at 56 weeks, the single test value will be used).

SECONDARY OUTCOMES:
Pediatric Eye Questionnaire (PedEyeQ) | 56 weeks
  Rasch scores for each questionnaire item will be obtained from published look-up tables available at www.pedig.net, and used to calculate a score for each participant and a separate treatment group mean for the three PedEyeQ domains of the Child, Proxy and Parent PedEyeQ at randomization and at each visit. Scores will also be converted to a 0-100 scale to aid in interpretation. Multiplicity adjusted two sided P-values and confidence intervals will be produced.
  Child PedEyeQ: Functional Vision, Bothered by Eyes and Vision, Social, Frustration / Worry Proxy PedEyeQ: Functional Vision, Bothered by Eyes and Vision, Social, Frustration / Worry, Eyecare Parent PedEyeQ: Impact on Parent and Family, Worry about Child's Eye Condition, Worry about Self-perception and Interactions, Worry about Functional Vision
Proportion Achieving Stable Resolved Outcome with Spectacles Alone | 56 Weeks
  The proportion of participants in the Sequential Spectacles group who achieve "stable resolved" outcome status with spectacles alone will be calculated, along with a multiplicity adjusted two sided P-value and confidence interval.
Proportion of participants who achieve Binary distance visual acuity outcomes | 56 weeks
  The proportion of participants who achieve the following binary outcomes will be tabulated by treatment group to aid in the interpretation of the primary outcome:
  * The proportion of participants with outcome amblyopic-eye distance VA improvement of ≥ 2 logMAR lines (≥ 10 letters if E-ETDRS) from baseline.
  * The proportion of participants with stable resolved VA.
  Poisson regression with the log link will be used to estimate the relative risk of each outcome for the sequential versus simultaneous and a multiplicity adjusted two sided P-value and confidence interval. The Poisson models will include an adjustment for baseline amblyopic eye VA.
  In the event the number of outcomes is too small for reliable estimation with Poisson regression,43 a treatment group difference and 95% confidence interval will be estimated using the Farrington-Manning Score test or other exact method with no adjustment for baseline VA.
Time to Stable Resolved Amblyopia | 56 weeks
  For those participants who are classified as "stable resolved," the time from baseline to the time meeting that classification will be compared between treatment groups, using a Kaplan-Meier analysis with the logrank test. Multiplicity adjusted two sided P-values and confidence intervals will be produced.
Difference in Mean Change of Distance Visual Acuity after 8 Weeks on Randomized Treatment | 56 Weeks
  An analysis of covariance (ANCOVA) will be performed to compute the difference in mean change in amblyopic-eye distance logMAR VA after 8 weeks between the sequential and simultaneous treatment groups, adjusted for baseline amblyopic eye distance VA, and a multiplicity adjusted two sided P-value and confidence interval will be constructed on the treatment group difference for each time point.
Change in binocularity levels | 56 Weeks
  Binocularity will be assessed on an ordered scale combining the results of the Randot Preschool Test, Randot butterfly, and Worth 4-Dot (W4D) at near. Results of each individual test also will be tabulated at baseline and at the final study visit according to treatment group.
  The possible levels of binocularity will be 40, 60, 100, 200, 400, 800 seconds of arc (Randot Preschool test), 2000 seconds of arc (Randot butterfly), binocular perception by W4D (4 or 5 lights), or no binocular perception by W4D (2 or 3 lights). This yields an ordered binocularity scale with 9 ordered levels. The change in binocularity levels for each test will be tabulated and compared between treatment groups using the exact Wilcoxon rank-sum test. The proportion of participants in each treatment group unable to perform testing will be tabulated but these participants will not be included in the analysis of change.
Difference in mean change in amblyopic-eye log contrast sensitivity | 56 weeks
  Contrast sensitivity scores range from unable (<0.90), and then from 0.90 to 2.05 (by 0.05 log contrast sensitivity units). An analysis of covariance (ANCOVA) will be performed to compute the difference in mean change in amblyopic-eye log contrast sensitivity units between the sequential and simultaneous treatment groups, adjusted for baseline amblyopic eye contrast sensitivity, and a multiplicity adjusted two sided P-value and confidence interval will be produced.

CONTACTS AND LOCATIONS:
Overall Officials: Vivian Manh, Study Chair — Seattle Children's Hospital, University of Washington; Michael Gray, Study Chair — Children's Hospital Medical Center, Cincinnati
Locations (68):
- United States (68):
  - UAB Pediatric Eye Care; Birmingham Health Care, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Midwestern University Eye Institute, Glendale, Arizona
  - Arizonia Pediatric Eye Specialists, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - Univ. of California- Berkeley, Berkeley, California
  - Marshall B. Ketchum University, Fullerton, California
  - Univ of California, Irvine- Gavin Herbert Eye Institute, Irvine, California
  - Loma Linda University Health Care, Dept. of Ophthalmology, Loma Linda, California
  - Children's Hospital of Los Angeles (CHLA), Los Angeles, California
  - Stanford University, Palo Alto, California
  - Western University College of Optometry, Pomona, California
  - University of California, Davis, Sacramento, California
  - University of California San Francisco Department of Ophthalmology, San Francisco, California
  - Eye Physicians & Surgeons, PC, Milford, Connecticut
  - Nova Southeastern University College of Optometry, The Eye Institute, Fort Lauderdale, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - University of South Florida (USF) Eye, Tampa, Florida
  - St Luke's Hospital, Boise, Idaho
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Ticho Eye Associates, Chicago Ridge, Illinois
  - Midwestern U Chicago College of Optometry, Downers Grove, Illinois
  - Progressive Eye Care, Lisle, Illinois
  - Indiana School of Optometry, Bloomington, Indiana
  - Indiana University School of Optometry, Indianapolis, Indiana
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - Wilmer Eye Institute, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Boston Children's Hospital Waltham, Boston, Massachusetts
  - Corewell Health, Grand Rapids, Michigan
  - Pediatric Ophthalmology, P.C., Grand Rapids, Michigan
  - Zenith Vision Development Center, Duluth, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - PineCone Vision Center, Sartell, Minnesota
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - St. Louis Children's Hospital Eye Center, St Louis, Missouri
  - U of MO St. Louis College of Optometry, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Ross Eye Institute, University of Buffalo, Med School Dept Ophthalmology, Buffalo, New York
  - NYU Langone Health, New York, New York
  - State University of New York, College of Optometry, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Eye Center, Durham, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Ohio State University College of Optometry, Columbus, Ohio
  - Dean A. McGee Eye Institute, Oklahoma City, Oklahoma
  - River View Family Eyecare, Albany, Oregon
  - Casey Eye Institute, Portland, Oregon
  - Pediatric Ophthalmology of Erie, Erie, Pennsylvania
  - Conestoga Eye, Lancaster, Pennsylvania
  - Wills Eye Hospital, Philadelphia, Pennsylvania
  - Salus University/Pennsylvania College of Optometry, Philadelphia, Pennsylvania
  - UPMC Children's Eye Center of Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Prisma Health, Columbia, South Carolina
  - Southern College of Optometry, Memphis, Tennessee
  - Vanderbilt University Medical Center - Vanderbilt Eye Institute, Nashville, Tennessee
  - Pediatric Eye Specialists, LLP, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - Texas Tech University Health Science Center, Lubbock, Texas
  - University of the Incarnate Word, San Antonio, Texas
  - San Antonio Eye Center, San Antonio, Texas
  - University of Incarnate Word Rosenberg School of Optometry, San Antonio, Texas
  - Rocky Mountain Eye Care Associates, Salt Lake City, Utah
  - Virginia Pediatric Eye Center, Norfolk, Virginia
  - Seattle Children's Hospital, University of Washington, Seattle, Washington
  - Spokane Eye Clinical Research, Spokane, Washington
  - Snowy Range Vision Center, Laramie, Wyoming

IPD SHARING:
Plan to Share IPD: Yes
In accordance with the NIH data sharing policy, a de-identified database is placed in the public domain on the Pediatric Eye Disease Investigator Group (PEDIG) public website after the completion of each protocol and publication of the primary manuscript.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available after publication.
Access Criteria: Users accessing the data must enter an email address.
URL: http://pedig.jaeb.org

DOCUMENTS (1):
  • Informed Consent Form (2020-07-22): https://cdn.clinicaltrials.gov/large-docs/90/NCT04378790/ICF_000.pdf